CLINICAL TRIAL: NCT02200952
Title: Luteal Phase Supplementation With Recombinant LH After GnRh Agonist Oocytes Triggering in Women at Risk of OHSS
Status: Completed | Type: Observational
Sponsor: San Carlo Public Hospital, Potenza, Italy (Other)
Responsible Party: Principal Investigator, Assunta Iuliano, MD, MD, PhD, San Carlo Public Hospital, Potenza, Italy
Other Study IDs: Luveris75UI
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS; Oocytes triggering; GnRh agonist triggering; Luteal phase supplementation; recombinant LH
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients at risk of OHSS: Patients at risk of OHSS on the oocytes triggering day with an oestradiol > 4000pg/ml or a number of follicles greater than 24 of a diameter greater than 12 mm
  Interventions: Drug: recombinant LH

INTERVENTIONS:
Drug: recombinant LH — recombinant LH twice/day for 10 days from pick up
  Other Names: Luveris rLH by Merck Serono

SUMMARY:
The purpose of this study is to prove that luteal phase supplementation with recombinant LH can solve the luteal phase deficiency after Gnrh agonist oocytes triggering in women at risk of OHSS

DETAILED DESCRIPTION:
The investigators enrolled patients, undergoing controlled ovarian stimulation for an IVF/ICSI cycles, who on the day of oocytes triggering were at risk of OHSS.

These patients had an estradiol > 4000 pg/ml and more than 24 follicles with a diameter greater than 12 mm.

The investigators used 0,2 mg of triptorelin for the oocytes triggering and supplemented the luteal phase with recombinant LH at a dose of 75 UI twice/day for 10 days and vaginal gel progesterone and oral oestradiol for 14 days The investigators measured bhCG at 14 days from the pick up. In case of positive bhCG we have defined the IVF/ICSI outcome: Pregnancy Rate and Implantation Rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with an oestradiol > 4000 pg/ml on the oocytes triggering day
* patient with more than 24 follicles of diameter greater than 12 mm on the oocytes triggering day

Exclusion Criteria:

* patients with no risk of OHSS on the oocytes triggering day
* patients with an oestradiol < 4000 pg/ml on the oocytes triggering day
* patient with less than 24 follicles of diameter greater than 12 mm on the oocytes triggering day

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients undergoing controlled ovarian hyperstimulation
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-06-30 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate and Implantation Rate | From 14 days after the pick up to six weeks of gestation
  We measured bhCG after 14 days from the pick up. In presence of a positive value of bhCG we evaluated IVF/ICSI outcome through the pregnancy rate and implantation rate.

SECONDARY OUTCOMES:
Ealy and Late Ovarian Hyperstimulation Syndrome | From 9 days after pick up to 12 weeks of gestation
  We evaluated early and late ovarian hyperstimulation syndrome according the practice committee of ASRM 2008 and Current Clinical Guideline for OHSS of 2010

CONTACTS AND LOCATIONS:
Overall Officials: Assunta Iuliano, MD, PhD, Principal Investigator — San Carlo Public Hospital, Potenza, Italy
Locations (1):
- San carlo Public Hospital, Potenza, Basilicate, Italy

REFERENCES:
- [Background] Papanikolaou EG, Verpoest W, Fatemi H, Tarlatzis B, Devroey P, Tournaye H. A novel method of luteal supplementation with recombinant luteinizing hormone when a gonadotropin-releasing hormone agonist is used instead of human chorionic gonadotropin for ovulation triggering: a randomized prospective proof of concept study. Fertil Steril. 2011 Mar 1;95(3):1174-7. doi: 10.1016/j.fertnstert.2010.09.023. Epub 2010 Oct 27. PMID 20979997